CLINICAL TRIAL: NCT03628378
Title: Outcomes in Free-hand Versus Sensor-guided Balancing in Total Knee Arthroplasty: a Randomized Controlled Trial
Brief Title: Orthosensor vs Conventional Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jeffrey Geller, Professor of Orthopaedic Surgery, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AAAR6137
Record Dates: First submitted 2018-07-26; First posted 2018-08-14 (Actual); Results first posted 2024-09-24 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Non-Sensor Group (No Intervention): Patients will undergo standard total knee replacement surgery without Verasense assisted balancing technology.
- Sensor Group (Experimental): Patients will undergo total knee replacement surgery with Verasense assisted balancing technology.
  Interventions: Device: Verasense

INTERVENTIONS:
Device: Verasense — Ligamentous balancing device
  Other Names: Orthosensor
  Arms: Sensor Group

SUMMARY:
In a randomized-controlled fashion, this investigation will evaluate the use of the Verasense technology to achieve optimal TKA balance. Patients will be randomized to either: 1) undergo manual soft tissue balancing or 2) soft tissue balancing with the Verasense. The primary outcomes of interest will include patient-reported outcomes as well knee range of motion at 3 months, 6 months, 1 year, and 2 years. Secondary outcomes of interest will include pain level as assessed by the visual analogue scale (VAS) in the acute post-operative and follow up periods, ambulation distance during inpatient physical therapy postoperatively, surgical time, tourniquet time, amount of opioid consumption, length of hospital stay, incidence of arthrofibrosis and subsequent manipulation under anesthesia. The investigators hypothesize that the use of the Verasense technology will lead to improved soft tissue balancing in TKA and ultimately result in favorable patient-reported outcomes and postoperative knee range of motion.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is one of the most successful surgical procedures performed worldwide, and if conducted properly, has proven to improve pain, knee range of motion, and ultimately quality of life. Approximately 700,000 TKAs are performed annually in the United States, and this number is projected to increase to 3.48 million annually by 2030. Unfortunately, roughly 20% of patients who undergo TKA are dissatisfied with their outcome and this number has remained stagnant for the past decade.Patient satisfaction after TKA is predominantly driven by postoperative pain and function.

Outcomes in TKA are influenced by multiple factors, stemming from patient-specific factors and surgically modifiable factors. Patient specific factors include body mass index (BMI), preoperative range of motion (ROM), psychological status, and other comorbidities; examples of surgically modifiable factors include the type of prosthesis utilized, posterior condylar offset, posterior tibial slope, and soft tissue balancing. Knee arthritis is a disease not only of the condylar surfaces, but of the soft tissues as well. As such, the success of a TKA depends on the ultimate restoration of the integrity of the knee articular surfaces,necessitating two critical elements, beginning with precise osteotomies and ending with soft tissue balancing to realign the lower extremity to a neutral mechanical axis.

In the last three decades, this first element has been addressed by major technological advances to perform precise and reproducible osteotomies, most recently with the development of computer-assisted navigation and validation techniques and modalities that allow osteotomies based on anatomical jigs created by CT imaging of the patient's knee.

Despite these advances, little advancement has been appreciated by the second element-soft tissue balancing.While precise osteotomies are critical to the success of a TKA, they do not address ligamentous stability and balance, which if absent, leads to knee instability, stiffness, accelerated prosthetic wear, aseptic loosening, and premature implant failure. Soft tissue imbalance accounts for 35% of early TKA revisions in the United States. Soft tissue balancing in TKA has traditionally been more of an art than a science, relying exclusively on the surgeon's subjective assessment based on nebulous tactile feedback after completion of the osteotomies. The diseased soft tissues (i.e. ligaments) may be lengthened, tightened, or released to achieve balance, range of motion, and functional stability. However, these methods are numerous, variable, and above all, highly subjective. The individual experience of the surgeon, including fellowship training and procedural volume play a role in their ability to balance a knee properly.

Typically, it is only after many years of experience does the surgeon develop the ability to accurately assess stability in varus, valgus, anterior and posterior planes.Objective balancing of soft tissues in TKA may contribute to a decrease in pain, improve function, patient satisfaction, and ultimately decrease the rate of revision. The need for the transformation of TKA soft tissue balancing from an art to a science has been realized by a technology that allows surgeons to objectively quantify ligament balance by offering real-time, evidence-based data during TKA. The Verasense (Orthosensor Inc., Dania, FL) is a disposable wireless device embedded with force sensors and inserted into the tibial component during the trialing phase of surgery after gross balancing, allowing real-time loading values in the medial and lateral compartments of the knee and fine-tuning of the end result by further soft tissue releases to improve balance and stability.

Balance in TKA is defined as stability in the sagittal plane and less than 15 pounds difference in the medial and lateral compartments of the knee. In a multicenter study, intraoperative sensors were utilized to define balance and to correlate it with improved clinical outcomes. TKAs that had undergone said balancing were compared to unbalanced TKAs, with results showing improved Knee Society Score (KSS) and Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) between balanced (172, 14.5 points) and unbalanced (145.3, 23.8 points), respectively. The authors concluded that a well-balanced TKA was the most significant contributing factor to improved postoperative outcomes.

Similarly, Chow et al. investigated six-month patient-reported outcomes in a small retrospective cohort study with short-term follow up of six months comparing sensor-assisted to non-sensor-assisted TKA balancing. They reported that the KSS, Oxford Knee Score, and knee range of motion was significantly higher in the sensor-assisted cohort and that the rate of arthrofibrosis was lower in the sensor-assisted group, however, not statistically significant.

Further, Geller et al. retrospectively compared the incidence of arthrofibrosis before and after the implementation of the Verasense technology to assist with ligament balancing and reported a 5% rate of arthrofibrosis prior to implementation versus 1.6% after. In this same report, median length of surgery was 83 minutes before implementation compared to 115 minutes after. The authors reported that while the implantation of the sensor increased operative time, this additional time does not have a clinical impact and that the benefits outweigh this potential increase in operative time. Multiple reports in the literature have suggested that a well-balanced TKA, which leads to increased activity levels may be part of a cascade effect, which ultimately results in higher patient-reported outcome scores.

Unfortunately, soft tissue balancing is one of the only remaining aspects of TKA that has not benefited from a consensus based on quantitative measures and objective data. As the economic environment changes in medicine, coupled with a five-fold increase in TKAs performed and the subsequent need for less experienced surgeons to perform TKAs, it is imperative that the traditional subjectivity once relied upon be replaced by more empirical and clinical data to construct a scientific consensus of what balance is. In so doing, clinical outcomes may be improved, with a resultant decrease in the rate of early revisions, and ultimately significant savings in healthcare expenditures.While the literature has demonstrated a clear advantage by technology like the Verasense, previous studies have predominantly been underpowered, with short-term follow up, and unstandardized TKAs, including surgical approach, prosthetic designs, manufacturer, and above all, not randomized and controlled.

ELIGIBILITY:
Inclusion Criteria:

* Primary total knee replacement

Exclusion Criteria:

* Revision knee surgery
* Prior knee surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2022-06-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Geller, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - NewYork-Presbyterian Lawrence Hospital, Bronxville, New York
  - Columbia University Irving Medical Center, New York, New York

REFERENCES:
- [Background] Kurtz S, Ong K, Lau E, Mowat F, Halpern M. Projections of primary and revision hip and knee arthroplasty in the United States from 2005 to 2030. J Bone Joint Surg Am. 2007 Apr;89(4):780-5. doi: 10.2106/JBJS.F.00222. PMID 17403800
- [Background] Chow JC, Breslauer L. The Use of Intraoperative Sensors Significantly Increases the Patient-Reported Rate of Improvement in Primary Total Knee Arthroplasty. Orthopedics. 2017 Jul 1;40(4):e648-e651. doi: 10.3928/01477447-20170503-01. Epub 2017 May 8. PMID 28481384
- [Background] Jacobs CA, Christensen CP, Karthikeyan T. Patient and intraoperative factors influencing satisfaction two to five years after primary total knee arthroplasty. J Arthroplasty. 2014 Aug;29(8):1576-9. doi: 10.1016/j.arth.2014.03.022. Epub 2014 Mar 28. PMID 24768544
- [Background] Judge A, Arden NK, Cooper C, Kassim Javaid M, Carr AJ, Field RE, Dieppe PA. Predictors of outcomes of total knee replacement surgery. Rheumatology (Oxford). 2012 Oct;51(10):1804-13. doi: 10.1093/rheumatology/kes075. Epub 2012 Apr 24. PMID 22532699
- [Background] Kim KW, Han JW, Cho HJ, Chang CB, Park JH, Lee JJ, Lee SB, Seong SC, Kim TK. Association between comorbid depression and osteoarthritis symptom severity in patients with knee osteoarthritis. J Bone Joint Surg Am. 2011 Mar 16;93(6):556-63. doi: 10.2106/JBJS.I.01344. PMID 21411706
- [Background] Camarata DA. Soft tissue balance in total knee arthroplasty with a force sensor. Orthop Clin North Am. 2014 Apr;45(2):175-84. doi: 10.1016/j.ocl.2013.12.001. Epub 2014 Feb 1. PMID 24684911
- [Background] Churchill JL, Khlopas A, Sultan AA, Harwin SF, Mont MA. Gap-Balancing versus Measured Resection Technique in Total Knee Arthroplasty: A Comparison Study. J Knee Surg. 2018 Jan;31(1):13-16. doi: 10.1055/s-0037-1608820. Epub 2017 Nov 27. PMID 29179222
- [Background] Krackow KA. Instability in total knee arthroplasty: loose as a goose. J Arthroplasty. 2003 Apr;18(3 Suppl 1):45-7. doi: 10.1054/arth.2003.50069. PMID 12730928
- [Background] Gustke KA, Golladay GJ, Roche MW, Elson LC, Anderson CR. A new method for defining balance: promising short-term clinical outcomes of sensor-guided TKA. J Arthroplasty. 2014 May;29(5):955-60. doi: 10.1016/j.arth.2013.10.020. Epub 2013 Oct 24. PMID 24269069
- [Background] Fehring TK, Odum S, Griffin WL, Mason JB, Nadaud M. Early failures in total knee arthroplasty. Clin Orthop Relat Res. 2001 Nov;(392):315-8. doi: 10.1097/00003086-200111000-00041. PMID 11716402
- [Background] Meneghini RM, Ziemba-Davis MM, Lovro LR, Ireland PH, Damer BM. Can Intraoperative Sensors Determine the "Target" Ligament Balance? Early Outcomes in Total Knee Arthroplasty. J Arthroplasty. 2016 Oct;31(10):2181-7. doi: 10.1016/j.arth.2016.03.046. Epub 2016 Apr 4. PMID 27155997
- [Background] Incavo SJ, Wild JJ, Coughlin KM, Beynnon BD. Early revision for component malrotation in total knee arthroplasty. Clin Orthop Relat Res. 2007 May;458:131-6. doi: 10.1097/BLO.0b013e3180332d97. PMID 17224835
- [Background] Walker PS, Meere PA, Bell CP. Effects of surgical variables in balancing of total knee replacements using an instrumented tibial trial. Knee. 2014 Jan;21(1):156-61. doi: 10.1016/j.knee.2013.09.002. Epub 2013 Sep 19. PMID 24103411
- [Background] Geller JA, Lakra A, Murtaugh T. The Use of Electronic Sensor Device to Augment Ligament Balancing Leads to a Lower Rate of Arthrofibrosis After Total Knee Arthroplasty. J Arthroplasty. 2017 May;32(5):1502-1504. doi: 10.1016/j.arth.2016.12.019. Epub 2016 Dec 24. PMID 28109758
- [Derived] Sarpong NO, Held MB, Grosso MJ, Herndon CL, Santos W, Lakra A, Shah RP, Cooper HJ, Geller JA. No Benefit to Sensor-guided Balancing Compared With Freehand Balancing in TKA: A Randomized Controlled Trial. Clin Orthop Relat Res. 2022 Aug 1;480(8):1535-1544. doi: 10.1097/CORR.0000000000002168. Epub 2022 Apr 7. PMID 35394462

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Non-Sensor Group | Sensor Group
Started | 67 | 63
Completed | 67 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Non-Sensor Group | Sensor Group | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (9) | 72 (8) | 71 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 50 | 97
  Male | 20 | 13 | 33
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 67 | 63 | 130
BMI [Mean (Standard Deviation); unit: kg/m2] | 29 (6) | 30 (6) | 29.5 (6)

OUTCOME MEASURES:

1. Primary Outcome: Average Score on the 12-Item Short Form Survey (SF-12) - Physical Component
Description: SF-12 is a patient-reported outcome measure assessing the impact of health on an individual's everyday life. The SF-12 is composed of a mental component score and a physical component score.
  The score range for each component is 0 to 100. Scores above 50 indicate a better-than-average health-related quality of life, while scores below 50 suggest below-average health.
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale
  3 months | 46 (8) | 43 (8)
  1 year | 45 (8) | 46 (6)
  2 years | 49 (6) | 47 (6)

2. Primary Outcome: Average Score on the 12-Item Short Form Survey (SF-12) - Mental Component
Description: as for outcome 1
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale
  3 months | 48 (5) | 48 (7)
  1 year | 46 (7) | 45 (7)
  2 years | 43 (7) | 43 (6)

3. Primary Outcome: Average Score on the WOMAC Functional (F) Limitation Subscale
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a 24-item patient-report questionnaire used to assess pain (score range 0-20), stiffness (score range 0-8), and functional limitation (score range 0-68). Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC-F score is derived as the sum of the 17 item scores in the pain domain. It will be normalized and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the Functional score and multiplying by 100.
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale
  3 months | 22 (17) | 28 (19)
  1 year | 21 (20) | 22 (21)
  2 years | 13 (19) | 16 (21)

4. Primary Outcome: Average Score on the WOMAC Stiffness (S) Subscale
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a 24-item patient-report questionnaire used to assess pain (score range 0-20), stiffness (score range 0-8), and functional limitation (score range 0-68). Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC-S score is derived as the sum of the 2 item scores in the pain domain. It will be normalized and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the Functional score and multiplying by 100.
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale
  3 months | 35 (22) | 37 (19)
  1 year | 31 (21) | 30 (26)
  2 years | 18 (22) | 20 (27)

5. Primary Outcome: Average Score on the WOMAC Pain (P) Subscale
Description: The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is a 24-item patient-report questionnaire used to assess pain (score range 0-20), stiffness (score range 0-8), and functional limitation (score range 0-68). Higher scores indicate worse pain, stiffness, and functional limitations. The WOMAC-P score is derived as the sum of the 5 item scores in the pain domain. It will be normalized and expressed on a 0-100 scale. This is done by dividing raw score by the highest possible value of the Pain score and multiplying by 100.
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale
  3 months | 18 (15) | 25 (21)
  1 year | 16 (21) | 16 (18)
  2 years | 12 (17) | 12 (19)

6. Primary Outcome: Knee Society Functional Score (KSFS)
Description: The investigators will ask participants to answer survey questions about knee functionality on a scale of 0-100, 0 being the least functionality and 100 being the most functionality.
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale
  3 months | 68 (18) | 55 (21)
  1 year | 65 (22) | 68 (20)
  2 years | 77 (23) | 71 (26)

7. Primary Outcome: Average Arc of Range of Motion (Extension to Flexion)
Description: A normal range of motion is 0º extension (completely straight leg) to 130º (a fully flexed leg).
Time Frame: 3 months, 1 year, 2 years
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
degrees
  3 months | 116 (13) | 113 (11)
  1 year | 117 (13) | 119 (13)
  2 years | 117 (12) | 116 (12)

8. Secondary Outcome: Visual Analogue Scale Pain Level
Description: Pain levels on a scale from 1-10 (1 being the least amount of pain possible and 10 being the most amount of pain possible).
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
score on a scale | 3.2 (1.9) | 3.2 (1.7)

9. Secondary Outcome: Ambulation (Distance)
Description: ambulation distance during inpatient physical therapy (PT) postoperatively - presented in daily PT performance in feet.
Time Frame: 1 week
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Non-Sensor Group | Sensor Group
Number analyzed (Participants) | 67 | 63
feet | 351 (290) | 361 (263)

ADVERSE EVENTS:
Time Frame: Up to 2 years for study-specific parameters, such as periprosthetic joint infection (PJI), superficial wound drainage and arthrofibrosis.
Arm/Group | Non-Sensor Group | Sensor Group
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/63
Other Adverse Events (participants affected / at risk) | 0/67 | 0/63

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-14): https://cdn.clinicaltrials.gov/large-docs/78/NCT03628378/Prot_SAP_000.pdf